CLINICAL TRIAL: NCT04097912
Title: Persistence and Adherence to Low-Dose Aspirin for Primary and Secondary Prevention of Cardiovascular DiseasE Using OHDSI
Brief Title: Study to Gather Information to What Extent Patients Follow the Treatment Regimen of Low-dose Aspirin for Primary and Secondary Prevention of Diseases of the Heart and Blood Vessels
Acronym: PALACE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20749
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Myocardial Infarction; Stroke (Including Ischaemic Stroke and Transient Ischaemic Attack); Unstable Angina; Angina; Ischaemic Heart Disease
MeSH Terms: conditions — Myocardial Infarction; Stroke; Ischemic Attack, Transient; Angina, Unstable; Angina Pectoris; Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Low-dose aspirin users: Patients who receive low-dose aspirin (75-100mg) for either the primary or secondary prevention of cardiovascular disease (CVD).
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — 75-100mg

SUMMARY:
This study aims to gather information to what extent patients follow the treatment regimen of low-dose aspirin for primary and secondary prevention of diseases of the heart and blood vessels. Researcher will collect information about the percentage of time a patient has access to the medication, how long patients continue with the medication and of the proportion of patients who switch from dual-antiplatelet therapy (including low-dose aspirin) to a single antiplatelet therapy. The study will make use of secondary healthcare data sources converted in to Observational Medical Outcomes Partnership (OMOP) common data model within the Observational Health Data Sciences and Informatics (OHDSI) network.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Patients will be selected if they have at least two prescriptions for low-dose aspirin (75-100 mg) between 2008 and 2018 for either:

  * Primary prevention of CVD This is defined as patients who have no history of CVD any time prior to initiation of low-dose aspirin treatment are presumed to use for primary CVD prevention
  * Secondary prevention of CVD This is defined as patients who have a history of CVD any time prior to initiation of low-dose aspirin treatment
* Patients with at least two prescriptions of low-dose aspirin with a dosage of 75-100mg within the first year of the index date.
* Restricted to patients with observation for at least 12 months before and 12 after the index date.

Exclusion Criteria:

- Prescription of low-dose aspirin in 12 months before the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population included in the study cohort will consist of patients who receive low-dose aspirin (75-100mg) for either the primary or secondary prevention of CVD.
  For those being treated with low-dose aspirin for primary CVD prevention, no previous CVD events must have occurred any time prior to initiation of low-dose aspirin treatment. CVD events consist of myocardial infarction, stroke (including ischaemic stroke and transient ischaemic attack), unstable angina, angina, and ischaemic heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Adherence to low-dose aspirin | Retrospective analysis from 2007 to 2018
  Adherence low-dose aspirin use will be represented by the medication possession ratio (MPR)
Persistence to low-dose aspirin | Retrospective analysis from 2007 to 2018
  In terms of continuation and discontinuation:
  * Continuation at 30 and 60 day gaps
  * Discontinuation:
  * If patients switched to another antiplatelet therapy
  * If patients reinitiated low-dose aspirin >30 days and >60 days after end of supply i.e. of the pre-specified gap was exceeded
  * If patients stopped low-dose aspirin therapy completely

SECONDARY OUTCOMES:
Time to switch from dual-antiplatelet to a monotherapy | Retrospective analysis from 2007 to 2018

CONTACTS AND LOCATIONS:
Locations (2):
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.